CLINICAL TRIAL: NCT00366912
Title: Unloading Respiratory Muscles During NIV: Comparison of a Spontaneous and Auto-adjusting Controlled Mode
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer recruiting: participants are no longer being recruited or enrolled
Sponsor: Krankenhaus Kloster Grafschaft (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Aladin 2006
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Failure
Keywords: work of breathing; pressure time product; muscle pressures
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

INTERVENTIONS:
Device: non-invasive ventilation

SUMMARY:
Measurement of Work of breathing (WOB), as well as pressure time product (PTP) of transdiaphragmatic pressures to evaluate the degree of muscle activity and muscle unloading during non-invasive ventilation.

The study makes comparison of a new developed auto adjusting controlled mode and a regular spontaneous mode.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) reduces carbon dioxide in hypercapnic respiratory failure by unloading the respiratory muscles. Spontaneous modes of NIV are usually being used in these situations. Spontaneous modes have the disadvantage, that the patient has to trigger the ventilator. The work to activate the trigger (WT) is estimated to be as high as up to 50% of the total work of breathing dependent on the underlying disease. Elimination of WT would increase the degree of respiratory muscle unloading.

A new pressure controlled mode incorporated into the ventilogic mechanical ventilator (Weinmann, Germany) is capable of self adjusting respiratory parameters in a preset range according to the patient requirements.

After a short period where the patients spontaneous respiratory parameters are being analyzed, the ventilator slowly implements a pressure controlled mode that matches the patients requirements.

This study intends to investigate if this new mode achieves a higher degree of respiratory muscle unloading compared to a spontaneous mode.

ELIGIBILITY:
Inclusion Criteria:

* Healthy voluntary individuals
* PFT within normal limits

Exclusion Criteria:

* Disease of the upper GI-tract
* Any form of lung disease or disease of the upper airways
* Any form of muscular disease, especially neuromuscular disease pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Work of breathing, pressure time product

SECONDARY OUTCOMES:
comfort

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dellweg, M.D., Principal Investigator — Fachkrankenhaus Kloster Grafschaft
Locations (1):
- Fachkrankenhaus Kloster Grafschaft, Schmallenberg, North Rhine-Westphalia, Germany